CLINICAL TRIAL: NCT00660777
Title: Effects of OroPharyngeal Exercises on Patients With Moderate Obstructive Sleep Apnea: A Randomized, Controlled Study
Brief Title: Effects of OroPharyngeal Exercises on Patients With Moderate Obstructive Sleep Apnea
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Geraldo Lorenzi-Filho, Heart Institute (InCor) - University of Sao Paulo Medical School
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OPE-OSA
Record Dates: First submitted 2008-04-07; First posted 2008-04-17 (Estimated); Last update posted 2008-04-17 (Estimated); Status verified 2008-04

CONDITIONS: Obstructive Sleep Apnea
Keywords: oropharyngeal exercises; obstructive sleep apnea; speech therapy
MeSH Terms: conditions — Sleep Apnea, Obstructive; Communication Disorders | interventions — Nasal Lavage

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Sham Comparator): Control Group
  Interventions: Behavioral: Deep breathing, bilateral alternate chewing, nasal lavage
- 2 (Active Comparator): Therapy Group
  Interventions: Behavioral: Oropharyngeal exercises

INTERVENTIONS:
Behavioral: Deep breathing, bilateral alternate chewing, nasal lavage — Deep breathing, bilateral alternate chewing, nasal lavage
  Arms: 1
Behavioral: Oropharyngeal exercises — Oropharyngeal exercises (derived from speech language pathology) to the soft palate, tongue and facial muscles exercises as well as stomatognathic functions.
  Arms: 2

SUMMARY:
Background: Upper airway muscle weakness plays an important role in the genesis of obstructive sleep apnea (OSA). Oropharyngeal exercises are derived from speech therapy consisting of isometric and isotonic exercises directed to tongue, soft palate and lateral pharyngeal wall. We hypothesized that oropharyngeal exercises will attenuate OSA severity.

We will include 30 moderate OSA patients (apnea-hypopnea index (AHI), between 15 and 30 events/hour) that will randomize to 3 months of general measurements and daily nasal lavage (n=15, control) or daily oropharyngeal exercises (~30 min) plus nasal lavage (n=16). Full polysomnography, anthropometric measurements, questionnaires derived from Berlin, Epworth and Pittsburgh evaluating quantitatively (range) snoring frequency (0-4) and intensity (1-3), daytime sleepiness (0-24) and sleep quality (0-21), respectively will be performed at baseline and study end.

DETAILED DESCRIPTION:
Patients: Eligible patients aged between 25 e 65 years old with a recent diagnosis of moderate OSA evaluated in the sleep laboratory, Pulmonary Division, Heart Institute (InCor). We will exclude patients with one or more of the follow conditions: body mass index (BMI) >40 kg/m2; facial malformations; regular use of hypnotic medications, hypothyroidism, previous stroke, neuromuscular disease, heart failure, coronary disease, and severe obstructive nasal disease.

Polysomnography: All patients will be evaluated by full polysomnography. The person who analyzed the sleep study will be blind to the group allocation.

Questionnaire: We will employ questionnaires previously validated and used in Brazil: Snoring frequency (derived from the Berlin questionnaire); subjective daytime sleepiness (Epworth questionnaire); quality of sleep (Pittsburgh sleep quality questionnaire).

Control Group: Sham therapy will consisted of a weekly supervised section (~30 min) of deep breathing, through the nose, while sitting, followed by a practice of bilateral alternate chewing. The patients will be instructed to perform the same procedure at home once a day (30 min), plus alternate bilateral chewing and nasal lavage with application of 10 ml of saline in each nostril three times a day.

Study Group: The same schedule and set of instructions will be applied to the control group was given to these patients. Oropharyngeal exercises are derived from speech language pathology and include soft palate, tongue and facial muscles exercises as well as stomatognathic function exercises.

Experimental Design: After fulfilling entry criteria, the patients will be randomized for 3 months of control or treatment group, with oropharyngeal exercises. All patients will be evaluated by the speech language pathologist once a week for 30 minutes. Patients that failed to return for 3 consecutive weeks or failed to comply to the exercises schedule at home were excluded from the study. Polysomnography and questionnaires will be performed at the beginning and at the end of the study.

Primary outcome: Apnea-hypopnea index.

Secondary outcomes: Lowest oxygen saturation and sleep related questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 25 and 65 years old with a recent diagnosis of moderate obstructive sleep apnea

Exclusion Criteria:

* Body mass index (BMI) >40 kg/m2
* Facial malformations
* Regular use of hypnotic medications
* Hypothyroidism
* Previous stroke
* Neuromuscular disease
* Heart failure
* Coronary disease
* Severe obstructive nasal disease

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2004-02; Primary Completion 2007-10 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Apnea-hypopnea index | 3 months

SECONDARY OUTCOMES:
Lowest oxygen saturation | 3 months
Sleep related questionnaires | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Kátia Guimaraes, Principal Investigator — Heart Institute (InCor); Geraldo Lorenzi-Filho, MD, PhD, Principal Investigator — Heart Institute (InCor)
Locations (1):
- Heart Institute (InCor), São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Guimaraes KC, Drager LF, Genta PR, Marcondes BF, Lorenzi-Filho G. Effects of oropharyngeal exercises on patients with moderate obstructive sleep apnea syndrome. Am J Respir Crit Care Med. 2009 May 15;179(10):962-6. doi: 10.1164/rccm.200806-981OC. Epub 2009 Feb 20. PMID 19234106